CLINICAL TRIAL: NCT02147509
Title: Evaluation of the Therapeutic Effect of Bandage Contact Lenses on Dry Eye Caused by Sjogren's Syndrome
Brief Title: Evaluation of Therapeutic Effect of Bandage Contact Lenses ( BCL) on Dry Eye Caused by Sjogren's Syndrome
Acronym: BCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinyang Li (Other)
Responsible Party: Sponsor-Investigator, Jinyang Li, Eye Hospital, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BCL-018-SS
Record Dates: First submitted 2014-05-13; First posted 2014-05-26 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Sjögren's Syndrome Patients With Severe Dry Eye
Keywords: Dry eye; Therapeutic bandage contact lenses; The quality of life
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Severe dry eye (Experimental): 1. 0.02% Fm, SH
  2. 0.02% Fm, SH, AS
  3. 0.02% Fm, SH, 0.05% CsA
  4. 0.02% Fm, SH, tBCL (0.05% CsA: 0.05% cyclosporin A; tBCL: therapeutic bandage contact lenses; 0.02% Fm: 0.02% Fluorometholone; AS: Autologous Serum; SH: Sodium Hyaluronate)
  Interventions: Drug: 0.02% Fm, SH; Drug: 0.02% Fm, SH, 0.05% CsA; Other: 0.02% Fm, SH, tBCL; Drug: 0.02% Fm, SH, AS

INTERVENTIONS:
Drug: 0.02% Fm, SH — Sjogren's Syndrome patients with severe dry eye
  Other Names: baseline treatment
Drug: 0.02% Fm, SH, 0.05% CsA — Sjogren's Syndrome patients with severe dry eye
  Other Names: immunosuppression treatment
Other: 0.02% Fm, SH, tBCL — Sjogren's Syndrome patients with severe dry eye
  Other Names: BCL treatment
Drug: 0.02% Fm, SH, AS — Sjogren's Syndrome patients with severe dry eye
  Other Names: Autologous Serum Treatment

SUMMARY:
The purpose of this study is to evaluate the therapeutic effect and safety of therapeutic bandage contact lenses treating dry eye caused by Sjögren's syndrome.

DETAILED DESCRIPTION:
Comparisons were made between Sjögren's syndrome patients with severe dry eye on the subjective and objective therapeutic effects of the overnight therapeutic bandage contact lenses at different period (i.e. before wearing, after wearing 3 weeks, after another 3 weeks with new lens and after 6 weeks without wearing ) based on the results of examinations.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female between 18~70 years old without wearing contact lens.
* Diagnosis and classification: all patients should have the symptoms and signs of severe dry eye (conforming to grade 3 or 4 in DEWS2007). Should have at least two positive symptoms such as dryness, foreign body sensation, burning, asthenopia, red eye or secretion. Tear film breakup time (TFBUT) shorter than 5 seconds and/or Schirmer I less than 5 mm/5 min. Corneal fluorescein staining more than 6 scores and (or) more than 3 scores of bulbar conjunctiva lissamine green liquor.
* Both eyes of all patients were preliminarily examined, the patients with single eye that meets the criterion were also investigated. Objective indicators were investigated on each eye. While the ocular surface disease index (OSDI) scores and SF-36 results were evaluated on an individual base.
* All patients should not participate in other medical tests in the past 2 weeks.
* Should either not be treated with other medicine at present, or have been treated with other medicine but had paused more than 2 weeks

Exclusion Criteria:

* Pregnant or maternity: exclude the patients who are or will be pregnant or during breast feeding.
* Other surface diseases: exclude the patients who are suspected or complicated by other obvious ocular surface diseases.
* Severe systemic diseases: exclude the patients with severe primary diseases in heart, brain blood vessel, liver, kidney, hematopoietic system and so on.
* Intraocular surgery or trauma: exclude the patients with intraocular surgery or trauma during 6 months.
* Hormone replacement therapy : exclude post-menopausal women who are treated in hormone replacement therapy.
* Lacrimal punctum: exclude the patients who have been treated with lacrimal punctum in 1 month.
* Glaucoma or high IOP: exclude the patients who have glaucoma or high intraocular pressure (IOP) sores.
* Exclude the patients who are sensitive to steroid.
* Exclude the patients who can't wear the therapeutic bandage contact lens during the clinical study.
* Immunosuppressive therapies: exclude the patients who are using systemic steroid or immunosuppressive therapies which may influent the results of the evaluation of the therapeutic effect.
* Excluding the patients who may not be suitable for the clinical examination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
C Corneal fluorescein staining | up to 12 weeks
  Divide the corneal into 4 quadrants and score each quadrant:
  0 score-no stains
  1. score-between 1 and 3 spots stained
  2. scores-greater than or equal 4 spots stained
  3. scores-spots stained fusion or filamentary

SECONDARY OUTCOMES:
Visual acuity | up to 12 weeks
  statistical analysis by logMAR.
Tear film breakup time | up to 12 weeks
  The lower fornix was stained with fluorescein paper, after the patient blinked a couple of times, the length of time between the last blink and tear BUT was recorded in seconds using a biomicroscope with cobalt blue lightning
Schirmer I test | up to 12 weeks
  standard Schirmer paper (5 mm width x 35 mm length) was placed at the intersection point of the lateral and middle one-third quadrants of the lower eye lid without anesthesia,and the wetting level was recorded in mm after 5 minThe operation is completed in the same laboratory.
quality of the life | up to 12 weeks
  tested by The Medical Outcomes Study 36-Item Short-Form Health Survey
Symptom of the dryness | up to 12 weeks
  Tested by ocular surface disease index

OTHER OUTCOMES:
Bulbar conjunctiva lissamine green staining | up to 12 weeks
  Divide the bulbar conjunctiva into 3 quadrants and score each quadrant:
  0 score-no stain
  1. score-between 1 and 3 spots stained
  2. scores-greater than or equal 4 spots stained
  3. scores-spots stained fusion or filamentary

CONTACTS AND LOCATIONS:
Overall Officials: Jinyang Li, MD,PhD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Eye Hospital, Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Li J, Zhang X, Zheng Q, Zhu Y, Wang H, Ma H, Jhanji V, Chen W. Comparative Evaluation of Silicone Hydrogel Contact Lenses and Autologous Serum for Management of Sjogren Syndrome-Associated Dry Eye. Cornea. 2015 Sep;34(9):1072-8. doi: 10.1097/ICO.0000000000000515. PMID 26147835